CLINICAL TRIAL: NCT01285479
Title: The Multi-National Gilenya Pregnancy Exposure Registry in Multiple Sclerosis
Brief Title: The Gilenya Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CFTY720D2404
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Last update posted 2025-01-22 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: Fingolimod; FTY720; Gilenya; Multiple sclerosis; MS; Safety; Pregnancy; Pregnancy outcomes
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 23 Months

GROUPS / COHORTS (1):
- fingolimod: prescribed fingolimod 0.5 mg/day, including generic versions of fingolimod
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — fingolimod 0.5 mg/day, including generic versions of fingolimod

SUMMARY:
The purpose of the Multi-National Gilenya Pregnancy Exposure Registry in Multiple Sclerosis (MS) is to continuously monitor, evaluate, and assess for major and minor teratogenic effects in the offspring of women exposed to fingolimod before (up to 8 weeks before last menstrual period (LMP)) and during pregnancy in routine clinical practice. The overall aim is to collect and evaluate data on maternal, fetal, and infant outcomes and compare it with reference populations.

ELIGIBILITY:
Inclusion Criteria:

* Any woman with a diagnosis of MS
* Any woman currently pregnant
* Exposure to fingolimod during pregnancy or up to 8 weeks before LMP
* Signed informed consent

Exclusion Criteria:

* There are no specific exclusion criteria for this registry.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with MS who become pregnant and were exposed to at least one dose of Gilenya during pregnancy (or up to 8 weeks before last menstrual period).
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2011-10-15 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Frequency of major malformations associated with exposure to fingolimod during pregnancy | Up to 23 months
  Major malformations are defined as any structural defect with surgical, medical, or cosmetic importance recognized.
Frequency of minor congenital malformations associated to fingolimod during pregnancy | Up to 23 months
  Minor congenital malformations:
  * Minor anomalies, i.e., anomalies with no serious medical or cosmetic consequence to the child.
  * Positional deformities, i.e., a positional deformity that usually normalizes spontaneously after about 3 months of age, e.g., abnormal head shape, torticollis.
  * Features of pre-maturity.
  * Chromosome abnormalities.
  * Genetic disorders.

SECONDARY OUTCOMES:
Frequency of specific types of major and minor congenital malformations associated with exposure to fingolimod during pregnancy | Up to 23 months
  Frequency of specific types of major and minor congenital malformations associated with exposure to fingolimod during pregnancy would be collected
Number of spontaneous abortions, stillbirths and elective terminations; | Up to 23 months
  Number of spontaneous abortions, stillbirths and elective terminations will be collected to characterize the nature of pregnancy and other fetal outcomes associated with exposure to fingolimod during pregnancy
Number of occurrence of physical developmental delays as well as adverse effects on immune system development in infants around one year of age | Up to 23 months
  Number of occurrence of physical developmental delays as well as adverse effects on immune system development in infants around one year of age associated with exposure to fingolimod during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (61):
- United States (3):
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Cambridge, Massachusetts
  - Novartis Investigative Site, Grand Forks, North Dakota
- Argentina (2):
  - Novartis Investigative Site, Bahía Blanca, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Novartis Investigative Site, Box Hill, Victoria, Australia
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
- Belgium (2):
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro, Brazil
- Novartis Investigative Site, Saint-Laurent, Quebec, Canada
- Novartis Investigative Site, Bogotá, Colombia
- Novartis Investigative Site, Nicosia, Cyprus
- Novartis Investigative Site, Ostrava-Poruba, Czechia
- Denmark (4):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Sønderborg
- Finland (2):
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (2):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Cahors
- Novartis Investigative Site, Bochum, Germany
- Novartis Investigative Site, Athens, GR, Greece
- Hungary (2):
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Győr
- Novartis Investigative Site, Dublin, Ireland
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Italy (6):
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
- Novartis Investigative Site, Beirut, Lebanon
- Novartis Investigative Site, Mexico City, Mexico City, Mexico
- Novartis Investigative Site, Amsterdam, Netherlands
- Poland (2):
  - Novartis Investigative Site, Lubin
  - Novartis Investigative Site, Warsaw
- Portugal (2):
  - Novartis Investigative Site, Amadora
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Moscow, Russia
- Saudi Arabia (2):
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh
- Novartis Investigative Site, Bratislava, Slovak Republic, Slovakia
- Novartis Investigative Site, Maribor, Slovenia
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Gothenburg, Sweden
- Switzerland (4):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Sankt Gallen
- United Arab Emirates (2):
  - Novartis Investigative Site, Abu Dhabi
  - Novartis Investigative Site, Dubai
- United Kingdom (3):
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: https://www.gilenyapregnancyregistry.com — https://www.gilenyapregnancyregistry.com